CLINICAL TRIAL: NCT03181139
Title: Efficacy of Enhanced Recovery After Surgery Pathway for Total Mastectomy
Acronym: ERAS_Breast
Status: Completed | Type: Observational
Sponsor: Monica Harbell (Other)
Collaborators: Mount Zion Health Fund (Other)
Responsible Party: Sponsor-Investigator, Monica Harbell, Assistant Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Other Study IDs: ERASBreast
Record Dates: First submitted 2017-06-02; First posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Mastectomy; Breast Cancer Female
Keywords: Enhanced Recovery after Surgery (ERAS); Fast-track surgery; Pec Blocks; Mastectomy
MeSH Terms: interventions — Mastectomy, Simple

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pre-ERAS: Patients cared for prior to the implementation of the Enhanced Recovery after surgery for total mastectomy pathway
- post-ERAS: patients cared for after the implementation of the Enhanced Recovery after surgery for total mastectomy pathway. Pathway included preoperative acetaminophen and gabapentin, Pec blocks, multimodal analgesia postoperatively and aggressive PONV treatment.
  Interventions: Other: ERAS pathway for Total Mastectomy

INTERVENTIONS:
Other: ERAS pathway for Total Mastectomy — Enhanced Recovery after Surgery (ERAS) pathway for Total Mastectomy
  Groups: post-ERAS

SUMMARY:
Retrospective analysis of pre and post-Enhanced Recovery after Surgery for Total mastectomy pathway implementation.

DETAILED DESCRIPTION:
Retrospective analysis of pre- and post-Enhanced Recovery after surgery for total mastectomy pathway implementation in patients at Mount Zion Hospital. We examined perioperative opioid consumption, pain scores, post-operative nausea and vomiting, benzodiazepine use, length of stay for the time period before and after implementation of an Enhanced Recovery after Surgery pathway for Total mastectomy. Pathway features included preoperative acetaminophen and gabapentin, minimizing opioids, postoperative NSAIDs, Pecs blocks, and aggressive postoperative nausea and vomiting prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* female patients at least 18 years old undergoing total skin sparing mastectomy at University of California San Francisco Mount Zion hospital

Exclusion Criteria:

* patients undergoing concurrent bilateral salpingo-oophorectomy, flap reconstruction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients at UCSF Mount Zion hospital who were scheduled for total mastectomy
Sampling Method: Non-Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
perioperative opioid consumption | through study completion (average of 1 year)
  perioperative opioid consumption

SECONDARY OUTCOMES:
Post-operative nausea and vomiting (PONV) | through study completion (average of 1 year)
  incidence post-operative nausea and vomiting
postoperative benzodiazepine use | through study completion (average of 1 year)
  amount of benzodiazepines used postoperatively for treatment of muscle spasm
Length of stay (LOS) | through study completion (average of 1 year)
  Length of stay
Pain score | through study completion (average of 1 year)
  highest pain score perioperatively
Surgery duration | through study completion (average of 1 year)
  length of surgery (min)

IPD SHARING:
Plan to Share IPD: No